CLINICAL TRIAL: NCT05343247
Title: Evaluation of Dental Age of Children With Amelogenesis Imperfecta Using Cameriere European Formula and London Atlas
Brief Title: Dental Age Estimation by Different Methods in Patients With Amelogenesis Imperfecta
Status: Completed | Type: Observational
Sponsor: Istanbul University (Other)
Responsible Party: Principal Investigator, Yelda Kasımoğlu, Principal investigator, Istanbul University
Other Study IDs: 2021/76
Record Dates: First submitted 2022-04-18; First posted 2022-04-25 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2023-11

CONDITIONS: Amelogenesis Imperfecta; Dental Age Estimation
Keywords: children; dental age estimation; amelogenesis imperfecta; chronological age; London Atlas; Cameriere European Formula
MeSH Terms: conditions — Amelogenesis Imperfecta

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Children with AI
  Interventions: Diagnostic Test: Cameriere method; Diagnostic Test: London Atlas method
- Healthy controls with gender-age match
  Interventions: Diagnostic Test: Cameriere method; Diagnostic Test: London Atlas method

INTERVENTIONS:
Diagnostic Test: Cameriere method — Cameriere et al. designed a quantitative approach through a formula based on sex and the ratio between length and apex opening measurements of each lower left tooth.
Diagnostic Test: London Atlas method — The London Atlas requires the user to assess the tooth development and eruption and then match it to one of the 31 pictures of age categories.

SUMMARY:
The aim of this study is to investigate whether there is a significant difference in dental age between children with amelogenesis imperfecta (AI) and healthy controls using Cameriere European formula and London Atlas. If there is a significant difference in dental age between children with AI and healthy controls, it is aimed to create a new formula.

DETAILED DESCRIPTION:
One of the developmental enamel defects, amelogenesis imperfecta (AI), is also known as enamel hypoplasia/hypomineralization. It is a rare inherited disease that affects the enamel structure, amount and component in primary and permanent teeth, and it has been reported to be accompanied by some dental anomalies and nephrocalcinosis. Dental anomalies and nephrocalcinosis can affect tooth development, and there are limited studies examining tooth development in these individuals.Dental age is widely evaluated by pedodontists, forensic dentists and orthodontists. While a delay in tooth development may be associated with growth retardation and learning difficulties, dental age determination can also be used for forensic age determination for children whose birth information is uncertain. A clear assessment of maturation in children with continued growth is important in establishing a dental treatment plan.

Dental age is widely evaluated by pedodontists, forensic dentists and orthodontists. While a delay in tooth development may be associated with growth retardation and learning difficulties, dental age determination can also be used for forensic age determination for children whose birth information is uncertain. A clear assessment of maturation in children with continued growth is important in establishing a dental treatment plan.

There are two basic approaches to dental age determination in children:

1. evaluation of eruption of teeth in the oral cavity,
2. evaluation of the development and mineralization of crowns and roots on dental radiographs.

In many methods, the developmental stages of different numbers of permanent teeth are used.

One of the most widely used methods of dental age determination recently is the European formula of Cameriere et al., which is calculated based on open apex. It has been reported that this method has been tested on different population groups, and the results are accurate and reliable.

An atlas method was proposed by a group of London researchers in 2010. The Atlas shows all the teeth array images of certain age groups as a schematic series. Age determination is made by deciding which reference image matches the individual's panoramic radiography image more.

ELIGIBILITY:
Inclusion Criteria:

* 5-13 years old
* Healthy children
* Children with AI
* Patients without missing left mandibular permanent teeth on panoramic radiography

Exclusion Criteria:

* Children older than 5 years old and younger than 14 years (children that cannot be assessed by the Willems and Cameriere method)
* Poor quality panoramic radiography
* Patients who have received orthodontic treatment
* Patients who received restorative or endodontic treatment

Ages: 5 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study was conducted on gender-age matched healthy control group of children aged 5-13 years, who applied to Istanbul University Faculty of Dentistry, Department of Pedodontics, had an AI record in their anamnesis, had panoramic radiographs in the archive of the Department of Oral and Maxillofacial Radiology, Istanbul University Faculty of Dentistry.
Sampling Method: Probability Sample
Enrollment: 416 (Actual)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-04-15 (Actual); Study Completion 2024-04-23 (Actual)

PRIMARY OUTCOMES:
Correlation coefficient of London Atlas method. | day 1
  Dental age of children with AI and healthy controls assessed by the correlation coefficient.
Correlation coefficient of Cameriere European formula. | day 1
  Dental age of children with AI and healthy controls assessed by the correlation coefficient.

SECONDARY OUTCOMES:
Dental age estimation in children with AI | day 1
  Dental age estimation in Turkish children

CONTACTS AND LOCATIONS:
Locations (1):
- Istanbul University, Faculty of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No